CLINICAL TRIAL: NCT05988736
Title: Comparison Between McGrath and Macintosh Laryngoscopes for Double-lumen Tube Intubation in Patients Undergoing Thoracic Surgery, A Prospective Randomized Controlled Trial
Brief Title: Comparison Between McGrath and Macintosh Laryngoscopes for DLT Intubation in Thoracic Surgery Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Sadique Ali, Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-7215-21602
Record Dates: First submitted 2023-07-27; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Thoracic Diseases; Thoracic Neoplasms; Thoracic Empyema
MeSH Terms: conditions — Thoracic Diseases; Thoracic Neoplasms; Empyema, Pleural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Device: MaCintosh Laryngoscope (DL)
- Group B (Active Comparator)
  Interventions: Device: McGrath Laryngoscope (VL)

INTERVENTIONS:
Device: MaCintosh Laryngoscope (DL) — A conventional Laryngoscope. It is battery powered, with a detachable MaCintosh blade that contains a light source.
  Arms: Group A
Device: McGrath Laryngoscope (VL) — A video Laryngoscope that has a high-resolution video camera, and a light source at the cone end of the blade allowing for direct and indirect viewing of the glottis
  Arms: Group B

SUMMARY:
The goal of this RCT is to compare outcome with McGrath vs Macintosh laryngoscopes among patients undergoing thoracic surgery. The main questions it aims to answer are,

1. Rate of successful intubation at first attempt and
2. Time for intubation required with each device. Participants are required to sign the informed consent for, they will be placed in two groups, Group A: Macintosh (DL) Group B: McGrath (VL) Researchers will compare in Group A: Macintosh (DL) and Group B: McGrath (VL) the differences in rate of successful intubation at first attempt and time for intubation required with each device.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* American Society of Anaesthesiologists physical status (ASA) I, II, III
* Elective thoracic surgery patients, requiring one lung ventilation.

Exclusion Criteria:

* Patients requiring rapid sequence induction
* Patients with a structural problem in the airway on chest radiography
* History of difficult intubation
* Planned tracheostomy \ the presence of a tracheostomy

  * Patients with a BMI >35 kg\m2. Who at risk of regurgitation\ Aspiration
  * Anticipated Difficult Airway (Mallampati IV)
  * Pre-existing sore throat or hoarseness, or recent respiratory infection (<15 days)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Time required for correct placement of the Double Lumen Tube (DLT). | During intervention time period
  Time will be measured in seconds during laryngoscopy while placement of Double Lumen Tube (DLT) until appearance of end tidal carbon dioxide on capnograph.
Successful Intubation at first attempt. | immediately after Intervention.
  The number of times the laryngoscope will be inserted.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan